CLINICAL TRIAL: NCT00519337
Title: The Impact of Ascorbic Acid Therapy on Inflammatory Mediators in Cardiothoracic Surgery Patients: The Atrial Fibrillation Suppression Trial IV (AFIST IV) Pilot Study
Brief Title: Impact of Ascorbic Acid on Post-Cardiothoracic Surgery Inflammation
Acronym: AFIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: The Gustavus and Louise Pfeiffer Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WHIT002743HE
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Cardiac Surgery; Inflammation
Keywords: Atrial Fibrillation; cardiac surgery; ascorbic acid; vitamin-c; inflammation
MeSH Terms: conditions — Inflammation; Atrial Fibrillation | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ascorbic acid
  Interventions: Drug: Ascorbic acid
- 2 (Placebo Comparator): Identical placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic acid — Ascorbic acid, 2 g p.o. the night before surgery followed by 500mg B.I.D. for 4 post-operative days
  Other Names: Vitamin-C
  Arms: 1
Drug: Placebo — Placebo capsule, 4 capsules the night before surgery followed by 1 capsule B.I.D. for 4 postoperative days
  Other Names: Identical Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to see if ascorbic acid (Vitamin-C) therapy will reduce inflammation following heart surgery.

DETAILED DESCRIPTION:
Atrial Fibrillation is a significant cause of morbidity following cardiothoracic surgery. Despite prophylactic therapy with beta-blockers and amiodarone, post-operative atrial fibrillation occurs in approximately 22% of patients. We believe that by reducing the inflammation that is caused during CTS, we can see further improvements without any negative effects on hemodynamics. Ascorbic acid, a free radical scavenger has been found to lower inflammation mediators but never in a CTS population. This study will help determine the affect of ascorbic acid on the inflammation associated with CTS.

ELIGIBILITY:
Inclusion Criteria:

* Cardiothoracic surgery

Exclusion Criteria:

* Pregnancy
* Prior hypersensitivity to ascorbic acid
* Renal Calculi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
In CTS patients receiving standard of care therapy,evaluate the effect of ascorbic acid therapy on c-reactive protein (CRP) concentration on post-CTS day 3 and the total post-CTS systemic exposure to CRP over 4 days. | 4 Postoperative Days

SECONDARY OUTCOMES:
Evaluate the effect of high intensity versus low intensity statin therapy on blood concentrations of fibrinogen, and White blood cell count on post-CTS days 3 and the total post-CTS systemic exposure to these biomarkers over 4 days. | 4 Postoperative Days

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael White, Pharm.D., Principal Investigator — Hartford Hospital, University of Connecticut
Locations (1):
- Hartford Hosptial, Hartford, Connecticut, United States